CLINICAL TRIAL: NCT01627899
Title: One Touch VerioIQ US Clinical Outcomes Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Business decision to terminate trial
Sponsor: LifeScan (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 3091611
Record Dates: First submitted 2012-06-22; First posted 2012-06-26 (Estimated); Results first posted 2018-08-02 (Actual); Last update posted 2018-08-02 (Actual); Status verified 2018-07

CONDITIONS: Diabetes
Keywords: Blood glucose monitor; Pattern management; Pattern guide; Education
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- VerioIQ (Other): Subjects replaced own Blood Glucose Monitoring system with VerioIQ.
  Interventions: Device: One Touch VerioIQ Blood Glucose Monitor

INTERVENTIONS:
Device: One Touch VerioIQ Blood Glucose Monitor — BGM with pattern alert technology and with associated pattern guide

SUMMARY:
Evaluation of the clinical benefits of One Touch VerioIQ system

DETAILED DESCRIPTION:
Evaluation of the clinical benefits of the One Touch VerioIQ system. The system contains pattern alert technology and comes with educational material (Pattern guide) which provides additional support and insights to patients and health care providers to help them make more informed decisions during blood glucose management.

ELIGIBILITY:
Inclusion Criteria:

* male or female at least 18 to 80 years old
* ADA guidelines for FPG and PPG appropriate
* A1C greater or equal to 8.0% and less than or equal to 10.5%
* lab A1C greater than or equal to 8.0% in the last 6-12mths
* Diagnosed with type 1 or 2 in at least last 1 year
* on stable dose of OADs for at least 3mths prior to screening
* willingness to test 7 BGM tests per day
* willing to remain on same therapy as baseline (MDI) for duration of study

Exclusion Criteria:

* unlikely to be compliant to study procedures
* has or has currently used One Touch VerioIQ
* Is on fixed doses of insulin for MDI therapy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2012-10-01 (Actual); Primary Completion 2013-05-01 (Actual); Study Completion 2013-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Priscilla Hollander, MD, Principal Investigator — Baylor Endocrine Center, 3600 Gaston Avenue Wadley Tower, Suite 656, Dallas, TX 75246, Phone: 214-820-3466, Fax: 214-820-3468

RESULTS

PARTICIPANT FLOW:
Recruitment Details: At medical clinic.
Groups:
- OneTouch VerioIQ BGMS: Subjects replaced own Blood Glucose Monitoring system (BGMS) with OneTouch VerioIQ
Period: Overall Study
Arm/Group | OneTouch VerioIQ BGMS
Started | 5
Completed | 0
Not Completed | 5
Not completed — Study terminated early by sponsor. | 5

BASELINE CHARACTERISTICS:
Population: No data was analysed including demographics as study was terminated early before any data was collected.
Arm/Group | OneTouch VerioIQ BGMS
Number analyzed (Participants) | 5
Age, Customized [Count of Participants; unit: Participants] — Population: No data was analysed including demographics as study was terminated early before any data was collected.
  Participants
    Unknown | 5
Sex/Gender, Customized [Count of Participants; unit: Participants] — Population: No data was analysed including demographics as study was terminated early before any data was collected.
  Participants
    Unknown | 5

OUTCOME MEASURES:

1. Primary Outcome: Change in A1C From Baseline to Week 24
Description: Change in A1C from baseline to week 24
Time Frame: 24 weeks
Population: Study terminated early by sponsor, no analysis completed.
Arm/Group | OneTouch VerioIQ BGMS
Number analyzed (Participants) | 0

2. Secondary Outcome: Change in A1C From Baseline to Week 12
Description: Change in A1C from baseline to week 12
Time Frame: 12 weeks
Population: Study terminated early by sponsor, no analysis completed.
Arm/Group | OneTouch VerioIQ BGMS
Number analyzed (Participants) | 0

3. Secondary Outcome: Change in FPG From Baseline to 24 Weeks and Over Time
Description: Change in Fasting Plasma Glucose (FPG) from baseline to 24 weeks and over time
Time Frame: 24 weeks and over time
Population: Study terminated early by sponsor, no analysis completed.
Arm/Group | OneTouch VerioIQ BGMS
Number analyzed (Participants) | 0

4. Secondary Outcome: Change in Proportion of Subjects With A1C Less Than or Equal to 7.0% at Week 24
Time Frame: 24 weeks
Population: Study terminated early by sponsor, no analysis completed.
Arm/Group | OneTouch VerioIQ BGMS
Number analyzed (Participants) | 0

5. Secondary Outcome: Change in 30 Day Mean Glucose Comparing First Month to Last Month After 24 Weeks
Time Frame: 24 weeks
Population: Study terminated early by sponsor, no analysis completed.
Arm/Group | OneTouch VerioIQ BGMS
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | OneTouch VerioIQ BGMS
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

LIMITATIONS AND CAVEATS:
No data was analysed as study was terminated early before any data was collected.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No